CLINICAL TRIAL: NCT07117175
Title: A Clinical Study to Evaluate the Safety and Efficacy of Anti-human CD 7 CAR-NK Cell Injection in Subjects With Relapsed and Refractory CD7-positive Hematological Malignancy
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xianmin Song, MD, Professor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHSYXY-CAR-NK-CD7
Record Dates: First submitted 2025-08-04; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Immunology; Hematologic Malignancies; CAR-NK
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intravenous infusion of anti-human CD7 CAR-NK cell injection (Experimental): Infusion of anti-human CD7 CAR-NK cell injection at D0
  Interventions: Drug: Anti-human CD7 CAR-NK cell injection

INTERVENTIONS:
Drug: Anti-human CD7 CAR-NK cell injection — Administer anti-human CD7 CAR-NK cell injection on D0
  Other Names: CD7 CAR-NK cell injection

SUMMARY:
This study is a single-arm, open-label, dose-escalation clinical trial to explore the safety, tolerability, pharmacokinetics and pharmacodynamics characteristics of the drug; The efficacy of the study drug in subjects with relapsed/refractory CD7-positive hematological malignancies, and the expression of B cells, T cells, and NK cell subtypes in peripheral blood were preliminarily observed. At the same time, explporing the distribution of anti-human CD7 CAR-NK cells in tumor tissues after administration of anti-human CD7 CAR-NK cell injection, and evaluating the immunogenicity of anti-human CD7 CAR-NK cell injection . To evaluate the correlation between the proportion of CD7-positive tumor cells and the safety and efficacy of anti-human CD7 CAR-NK cell injection and the evaluation. To explore the pharmacokinetics (PK) and pharmacodynamics(PD) characteristics of bone marrow in Chinese medicine.

DETAILED DESCRIPTION:
"This study employed a dose escalation approach combining accelerated titration for the first dose group and the standard '3+3' rule for subsequent dose groups, aiming to minimize patient exposure to ineffective doses while reducing potential risks as much as possible. The study comprised three dose groups for single administration, with doses set at 1×10^7 CAR-NK cells/kg, 2×10^7 CAR-NK cells/kg, and 5×10^7 CAR-NK cells/kg. For the 1×10^7 CAR-NK cells/kg dose group, an accelerated titration method was applied: after obtaining informed consent, one eligible subject meeting the inclusion/exclusion criteria was enrolled into this group. A safety assessment was conducted 14-28 days after the first cell infusion. If no dose-limiting toxicity (DLT) occurred, the subject could proceed to the next dose group upon agreement between the investigator and sponsor. If DLT occurred in one subject, after evaluation by the investigator and sponsor, two additional subjects were enrolled into the same dose group for a 28-day observation period. If DLT events occurred in ≤1 of these three subjects, the study could advance to the next dose group; if DLT events occurred in >1 subject, the decision to continue was made through joint discussion between the investigator and sponsor.

Dose escalation to the 2×10^7 CAR-NK cells/kg dose group followed the standard '3+3' rule. This group initially enrolled three subjects. If no DLT occurred in all three subjects, the study could proceed to the 5×10^7 CAR-NK cells/kg dose group upon agreement between the investigator and sponsor. If one DLT occurred in this group, three additional subjects were enrolled for further observation of the same dose level. If the total number of DLT events among these six subjects was ≤1, the study could advance to the 5×10^7 CAR-NK cells/kg dose group with agreement. If more than one subject experienced DLT in this group, enrollment for this dose level was terminated, and the dose was reduced to complete enrollment of remaining subjects, as decided by the investigator and sponsor.

Dose escalation to the 5×10^7 CAR-NK cells/kg dose group also adhered to the standard '3+3' rule. This group first enrolled three subjects. After cell infusion, a 28-day safety assessment was completed. If no DLT occurred in all three subjects, the decision to continue dose escalation was made through joint discussion between the investigator and sponsor. If no further escalation was decided, the remaining subjects were enrolled in this dose group. If one DLT occurred among the first three subjects, three additional subjects were enrolled for further observation. If DLT events occurred in >1 of these six subjects, enrollment for this dose group was terminated, and the dose level was reduced to complete enrollment of remaining subjects.

If no maximum tolerated dose (MTD) was observed at the maximum dose of 5×10^7 CAR-NK cells/kg, the decision to add additional dose groups was made through joint discussion between the investigator and sponsor, with the new group still following the standard '3+3' rule. During the study, dose groups could be adjusted based on the tolerability, pharmacokinetics, pharmacodynamics, and efficacy of anti-human CD7 CAR-NK cells in patients, combined with prior CAR-NK treatment experience, as determined by the investigator and sponsor. This could involve adding or reducing groups or adjusting dose levels. If special safety or efficacy issues arose during dose escalation, the clinical study could be terminated after joint discussion between the investigator and sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years old, gender is not limited;
* The expected survival time exceeds 12 weeks;
* ECOG score 0 to 2 points;
* Comply with the 2022 WHO standards for acute myeloid leukemia (AML), lymphoblastic lymphoma/leukemia (LBL/ALL), and after testing, CD7-positive flow cytometry leukemia cells expressed CD7 by ≥70%; or immunohistochemical leukemia cells expressed CD7 ≥50%. At the same time, it meets the following relapse-refractory standards:

  1. Recurrence criteria: ≥5% of the original cells appear in the bone marrow after hematologic remission (except for the hematopoietic recovery period after chemotherapy); or 2 peripheral blood samples at least one week intervals; or extramedullary lesions appear. Patients with early relapse (recuring within 12 months after the first remission) can be directly enrolled, while patients with advanced relapse (recuring after the first remission) need to rescue at least one course of chemotherapy through the original effective induction regimen and no remission is achieved; all relapse patients should include selectable targeted drugs for at least one course of treatment without remission. Allogeneic hematopoietic stem cells recur after transplantation, no other effective treatment options are available, and there is no active acute graft-versus-host disease (GVHD) above 2 degrees.
  2. Refractory criteria: Complete remission was not achieved at the end of induction therapy, and complete remission was not achieved after second-line rescue chemotherapy or the treatment regimen containing optional targeted drugs. Patients with tumor burden exceeding 5%, patients with persistent micro-residual lesions (MRD) positive, or patients with extramedullary lesions are also considered eligible.
* The intravenous pathway required for collection can be established, without contraindications for white blood cell collection;
* Liver and kidney function and cardiopulmonary function meet the following requirements:

  1. Creatinine clearance (calculated by Cockcroft Gault formula) ≥60 mL/min or creatinine ≤2.5×ULN;
  2. The cardiac ejaculation fraction is greater than 50%, and there is no clinically significant electrocardiogram change;
  3. Baseline blood oxygen saturation is greater than 92%;
  4. Total bilirubin ≤3×ULN; ALT and AST ≤3×ULN;
* Be able to understand this test and have signed an informed consent form.

Exclusion Criteria:

* Use of immunosuppressive drugs or steroids within two weeks prior to cell collection, or the need for steroid or immunosuppressive drug use for more than two years.
* History of malignancy other than hematologic neoplasms within five years before screening, except for adequately treated cervical carcinoma in situ, basal cell, or squamous cell skin cancer, localized prostate cancer after curative surgery, ductal carcinoma in situ after curative surgery, and thyroid cancer after curative surgery;
* Active bacterial, viral, or fungal infections requiring treatment and not controlled; positive HBsAg or HBcAb (if positive, peripheral HBV-DNA testing is required with HBV DNA < detection limit to be eligible); positive HCV antibody with peripheral blood HCV RNA positivity; positive Treponema pallidum particle assay (TPPA); HIV antibody positivity;
* Inadequate function of major organs (cardiovascular system, lungs), active gastrointestinal bleeding within the past three months; uncontrolled hypertension or history of hypertensive crisis or hypertensive encephalopathy; significant cardiovascular risk history or evidence including any of the following: congestive heart failure, unstable angina pectoris, clinically significant arrhythmias (such as ventricular fibrillation, ventricular tachycardia); history of arterial thrombosis formation within the last three months (such as stroke, transient ischemic attack); symptomatic deep vein thrombosis or pulmonary embolism within six months prior to enrollment; previous coronary angioplasty procedure; cardioversion by electric shock; any clinically relevant complications that may pose a risk to the safety of the subject or interfere with study assessments, procedures, or completion;
* Any uncontrolled active disease that would preclude participation in the trial;
* Active and uncontrolled central nervous system involvement by disease process or a history thereof requiring treatment (e.g., epilepsy);
* Subjects receiving systemic corticosteroid therapy at screening who are expected to require long-term systemic corticosteroid therapy during the course of the study (inhaled and topical use excluded);
* Subjects who have used PD-1/PD-L1 monoclonal antibodies within three months prior to enrollment;
* Pregnant women and those lactating; subjects planning pregnancy within one year post-infusion or during/after treatment;
* Presence of uncontrollable active infection (simple urinary tract infection and upper respiratory tract infection excluded);
* Previous receipt of CAR-T/CAR-NK therapy or other genetically modified cellular therapies;
* Allogeneic transplant recipients without evident acute/chronic graft-versus-host disease and off immunosuppressive drugs for at least one month;
* Known allergy to any component of anti-human CD7 CAR-NK cell injection solution or chemotherapy regimen (cyclophosphamide and fludarabine);
* Any condition deemed by the investigator as likely to impair subject safety or interfere with study objectives; subjects considered unsuitable for this trial by investigators.
* Subjects unable to provide written informed consent due to illness affecting their ability to do so; unwillingness or inability to comply with study requirements.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-12-15 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity | Up to day 28
  To evaluate the incidence of DLT in patients with relapsed or refractory CD7-Positive Hematological Malignancies treated with anti-human CD7 CAR-NK cell injection, DLT is defined as any of the following events related to the study drug (including definitely related, probably related, and possibly related) that occurs within 14-28 days after the first dose of the investigational human CD7 CAR-NK cell injection (with appropriately extended observation duration for responders in dose groups showing therapeutic responses to assess whether DLT events resolve within the specified time frame), despite therapeutic interventions.
Incidence of adverse events | through study completion, an average of 2 year
  The occurence of study related adverse effects defined by NCI CTCAE5.0

SECONDARY OUTCOMES:
Evaluate the number of CAR-NK cells in subjects' peripheral blood | Through study completion, an average of 2 year
  Evaluate the number of Treg cells in subjects' peripheral blood after CD7 Car-NK cell injection administration
Analysis of the number changes of cytokine in peripheral blood. | Through study completion, an average of 2 year
  Analysis of the number changes of cytokine in peripheral blood,Levels of related cytokines (such as IL-6);
Analysis of the number changes of lymphocyte subsets in peripheral blood. | Through study completion, an average of 2 year
  Analysis of the number changes of lymphocyte subsets in peripheral blood, Including T/B/NK cells
Objective Response Rate (ORR) | Through study completion, an average of 2 year
  To evaluate the efficacy of CD7 Car-NK cell injection of relapsed or refractory CD7-Positive Hematological Malignancies subjects.
Duration of response after administration (DOR) | Through study completion, an average of 2 year
  Duration of response after administration (DOR),It refers to the time from the first assessment of CR or CRi or PR or MLFS to the first assessment of disease progression (Progressive Disease, PD) or death from any cause (including time post allogeneic hematopoietic stem cell transplantation).
Progression-free survival post-administration | Through study completion, an average of 2 year
  The time from cell infusion to the first assessment of tumor progression or death from any cause (including time post allogeneic hematopoietic stem cell transplantation).
Overall survival | Through study completion, an average of 2 year
  The time from the start of cell reinfusion to death due to any cause. For subjects who have dropped out before death, the last follow-up time will be recorded as the time of death.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No